

## Self-administered mindfulness interventions reduce stress in a large, randomized controlled multi-site study.

Alessandro Sparacio<sup>1,2</sup>, Hans IJzerman<sup>1,3</sup>, Ivan Ropovik<sup>4,5</sup>, Filippo Giorgini<sup>6</sup>, Christoph Spiessens<sup>7</sup>, [authors that contributed with the data collection with at least 70 participants], Gabriela M. Jiga-Boy<sup>2</sup>

<sup>1</sup>Université Grenoble Alpes, <sup>2</sup>Swansea University, <sup>3</sup>Institut Universitaire de France, <sup>4</sup>Charles University in Prague, <sup>5</sup>Presov University, <sup>6</sup>University of Milano-Bicocca, <sup>7</sup>Christoph Spiessens Coaching Solutions Ltd.

## PARTICIPANT INFORMATION SHEET

**Project title:** A large, multisite test of self-administered mindfulness

You are being invited to take part in some research. Before you decide whether or not to participate, it is important for you to understand why the research is being conducted and what it will involve. Please read the following information carefully.

What is the purpose of the research? We are conducting research on types of meditations that can be self-administered (that means, meditation exercises that you can do on your own, for example by using a smartphone application). We test the link between brief mindfulness exercises and how individuals feel after having done them. Your participation in this study will take approximately 25-30 minutes.

Who is carrying out the research? The project management team include Alessandro Sparacio (PhD student in the School of Psychology, Swansea University and Universite Grenoble Alpes, France), supervised by Dr Gabriela Jiga-Boy (School of Psychology, Swansea University), Dr Hans IJzerman (Université Grenoble Alpes & Institut Universitaire de France) and Dr Ivan Ropovik (Charles University in Prague & Presov University). Sites across the world will conduct data collection as well; their ethical applications will be submitted at their affiliated institutions, if requested.

**What happens if I agree to take part?** You will be randomly allocated to do an exercise that may or may not involve meditation. The experiment will be administered via the online platforms Qualtrics.

What do I need to do to take part? If you take part in this study, we ask you to <u>complete it via a smartphone</u> (not a computer!) and to <u>use your headphones during the entire study</u>. You will go through the following steps: First, we ask for your consent to take part. If you consent, you will be asked a series of brief questionnaires before the beginning of the experiment. Then you will be invited to participate in either a brief self-administered mindfulness session that will last 15 minutes or another exercise. At the end of the exercise, you will receive a short questionnaire measuring how you feel. Finally, we will ask for demographic information such as your age, gender identity, and your country of birth.

Are there any risks associated with taking part? The research has been approved by the School of Psychology, Swansea University Research Ethics Committee and by the Ethics Committee of the participating sites. There are no significant risks associated with participation. Some of the questions will ask you to report your emotions, and some of the exercises used involve mindfulness meditation. PLEASE DO NOT TAKE PART if you currently are or have been diagnosed with a mood disorder (for example: Major Depressive Disorder, Bipolar Mood Disorder, etc.) AND/OR if you have ever experienced psychosis episode(s). Thank you!

Data Protection and Confidentiality: Your data will be processed in accordance with the Data Protection Act 2018 and the General Data Protection Regulation 2016 (GDPR). All information collected about you will be kept strictly confidential. Your data will only be viewed by the research team. All electronic data will be stored on a Qualtrics account owned by Swansea University, UK. The servers are in the UK, not Australia. Data will then be downloaded from Qualtrics and will be stored as password-protected files on password-protected computers at Swansea University. Your consent information will be kept separately from your responses to minimise risk in the event of a data breach. Please note that the data we will collect for our study will be anonymous. The researchers will abide by local data protection laws when collecting personal data. When the research project is published your anonymised data will be uploaded to the Open Science Framework (OSF) webpage (https://osf.io/) and can be accessed by researchers outside of the current research team.

Please note that countries outside of the European Economic Area may not offer the same level of data privacy protection as in the UK. For sharing the information with researchers outside the EEA, we (the project management team) will abide by Swansea University's data protection and freedom of information regulations (http://www.swansea.ac.uk/the-university/world-class/vicechancellorsoffice/compliance-team/).

What will happen to the information I provide? An analysis of the information will form part of our report at the end of the study and may be presented to interested parties and published in scientific journals and related media. Note that all information presented in any reports or publications will be anonymous and unidentifiable.

**Is participation voluntary and what if I wish to later withdraw?** Your participation is entirely voluntary – you do not have to participate if you do not want to. If you decide to participate, but later wish to withdraw from the study, then you are free to withdraw at any time, without giving a reason and without penalty.

**Data Protection Privacy Notice.** The data controller for this project will be Swansea University, UK. The University Data Protection Officer provides oversight of university activities involving the processing of personal data, and can be contacted at the Vice Chancellor's Office.

Your personal data will be processed for the purposes outlined in this information sheet. Standard ethical procedures will involve you providing your consent to participate in this study by completing the consent form that has been provided to you or by ticking the box provided, if consent is collected with an online survey.

The legal basis that we will rely on to process your personal data states that processing is necessary for the performance of a task carried out in the public interest. This public interest justification is approved by the School of Psychology, Faculty of Medicine, Health and Life Science Research Ethics Committee, Swansea University.

The legal basis that we will rely on to process special categories of data states that processing is necessary for archiving purposes in the public interest, scientific or historical research purposes or statistical purposes.

How long will your information be held? Data will be preserved and accessible for a minimum of 10 years after completion of the research. Records from studies with major health, clinical, social, environmental or heritage importance, novel intervention, or studies which are on-going or controversial should be retained for at least 20 years after completion of the study. It may be appropriate to keep such study data permanently within the university, a national collection, or as required by the funder's data policy.

What are your rights? You have a right to access your personal information, to object to the processing of your personal information, to rectify, to erase, to restrict and to port your personal information. Please visit the Swansea University Data Protection webpages for further information in relation to your rights. Any requests or objections should be made in writing to the University Data Protection Officer: University Compliance Officer (FOI/DP), Vice-Chancellor's Office, Swansea University, Singleton Park, Swansea, SA2 8PP; Email: <a href="mailto:dataprotection@swansea.ac.uk">dataprotection@swansea.ac.uk</a>.

**How to make a complaint.** If you have any complaints or reservations about any ethical aspect of your participation in this research, you may contact the Committee through the Director, Research Ethics & Integrity (telephone (02) 9850 7854; email ethics@mq.edu.au). Any complaint you make will be treated in confidence and investigated, and you will be informed of the outcome.

What if I have other questions? If you have further questions about this study, please do not hesitate to contact us:



**Swansea** 

Alessandro Sparacio (PhD Student) School of Psychology, Swansea University Université Grenoble Alpes Email: 943633@swansea.ac.uk

Dr Gabriela Jiga-Boy (Supervisor) Senior lecturer School of Psychology, Swansea University Email: g\_jiga@swansea.ac.uk

## **Participant Consent Form**

Project title: A large, multisite test of self-administered mindfulness.

Name & Contact details of the principal researchers: Sparacio Alessandro, School of Psychology, Swansea University & Université Grenoble Alpes, Email: <u>943633@swansea.ac.uk</u>. <u>Dr</u> Gabriela Jiga-Boy, Senior lecturer, School of Psychology, Swansea University, UK; Email: <u>g.jiga@swansea.ac.uk</u>.

| | Participant initial |
|---|---|
| 1. I (the participant) confirm that I have read and understand the information sheet for the above study (dated:) which is attached to this form. | |
| 2. I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reasons. | |
| 3. I understand what my role will be in this research, and all my questions have been answered to my satisfaction by the information provided on the Participant Information Sheet provided. | |
| 4. I understand that I am free to ask any questions at the end of the study and I have been provided with the researchers' contact details. | |
| 5. I have been informed that the information I provide will be safeguarded. | |
| 6. I am happy for the information I provide to be used (anonymously) in academic papers and other formal research outputs. | |
| 7. I have been provided with the opportunity to download a copy of the Participant Information Sheet or to ask for one from the study researchers. | |
| 8. I agree to the researchers processing my personal data in accordance with the aims of the study described in the Participant Information Sheet. | |
| 9. I confirm that I am 18 years or older. | |

If you agree with all statements listed above, click YES.

If you disagree with any of the statements above, click **NO** and you will be taken to the end of this survey.

This study is being conducted by School of Psychology, Faculty of Medicine, Health and Life Science, Swansea University.

Thank you for your participation in this study! Your help is very much appreciated.